CLINICAL TRIAL: NCT01626651
Title: An Open-Label, Sequential Design Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Ibrutinib in Healthy Subjects
Brief Title: A Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of Ibrutinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100870; PCI-32765CLL1002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-06-18; First posted 2012-06-25 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Healthy; Ketoconazole; Ibrutinib
MeSH Terms: interventions — ibrutinib; Ketoconazole

ARMS (1):
- Ibrutinib and Ketoconazole (Experimental)
  Interventions: Drug: Ibrutinib; Drug: Ketoconazole

INTERVENTIONS:
Drug: Ibrutinib — A single oral dose of 120 mg ibrutinib (3 x 40 mg capsules) on Day 1, and 40 mg (1x 40 mg capsule) ibrutinib on Day 7.
Drug: Ketoconazole — Ketoconazole (400 mg [2 x 200 mg] once daily) will be orally administered on Days 4, 5, 6, 7, 8 and 9.

SUMMARY:
The purpose of this study is to assess the potential effects of ketoconazole on the pharmacokinetics of ibrutinib in healthy participants.

DETAILED DESCRIPTION:
This is a single-center, open-label (all people know the identity of the intervention), sequential design study in healthy men. All participants will receive ibrutinib on Day 1 and ibrutinib in combination with ketoconazole on Day 7. Food will be restricted from the evening before dosing until 4 hours after dosing on Days 1 and 7. Following an overnight fast, ketoconazole will be given on Days 4 to 6, 1 hour prior to ibrutinib dosing on Day 7, and again on Days 8 and 9. All ibrutinib and ketoconazole doses will be administered with water. The participants will leave the study center on Day 10.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kg/m2, and body weight not less than 50 kg
* Blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic
* Non-smoker
* Must agree to use an adequate contraception method during the study and minimally 3 months after the last dose of ibrutinib, and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Signed an informed consent document

Exclusion Criteria:

* History of or current clinically significant medical illness
* Clinically significant abnormal physical examination, vital signs or electrocardiogram (ECG)
* Clinically significant abnormal values for laboratorial tests
* Use of any prescription or nonprescription medication, except for acetaminophen, within 3 days before the first dose of the study drug is schedule
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 2 years

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Ibrutinib plasma concentrations after administration on Day 1 | over 72 hours after dosing on Day 1
Ibrutinib plasma concentrations after administration on Day 7 | over 72 hours after dosing on Day 7
Metabolite PCI-45227 plasma concentrations after administration on Day 1 | over 72 hours after dosing on Day 1
Metabolite PCI-45227 plasma concentrations after administration on Day 7 | over 72 hours after dosing on Day 7

SECONDARY OUTCOMES:
Ibrutinib urine concentrations after administration on Day 1 | over 72 hours after dosing on Day 1
Ibrutinib urine concentrations after administration on Day 7 | over 72 hours after dosing on Day 7
Metabolite PCI-45227 urine concentrations after administration on Day 1 | over 72 hours after dosing on Day 1
Metabolite PCI-45227 urine concentrations after administration on Day 7 | over 72 hours after dosing on Day 7
Incidence of adverse events as a measure of safety and tolerability | Approximately 41 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Neptune City, New Jersey, United States